CLINICAL TRIAL: NCT05964842
Title: Using Short Message Service Reminders, Phone Calls and Mobile Money Incentives to Enhance Linkage to Care of Presumptive Tuberculosis Patients in Uganda: a Randomised Controlled Trial
Brief Title: Using SMS Reminders, Phone Calls and Money Incentives to Enhance Linkage to Care of Presumptive TB Patients in Uganda
Acronym: MILEAGE4TB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: MILEAGE4TB
Record Dates: First submitted 2023-06-04; First posted 2023-07-28 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Presumptive TB; Loss to follow-up; SMS; Phone call; Cash incentives; Mobile health (mHealth); Pre-treatment loss to follow-up; Pre-diagnosis loss to follow-up
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: This will be an individual randomized controlled trial with five arms. The study arms will include; i) Standard of care (SOC - control group) ii) SMS only iii) phone call only iv) SMS and mobile money incentive v) Phone call and mobile money incentive
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Due to the nature of the intervention, participants will not be blinded to the study arm though data analysis will be blindly conducted.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Standard of care (Control) (No Intervention): Patients in this arm will receive the routine TB care, according to the Uganda Ministry of Health guidelines, that is; i) Patient screened for TB ii) Patient identified as presumptive and registered in the presumptive TB register iii) Patient referred for TB testing iv) Patient expected to return and pick results on their own drive vi) Positive TB patients initiated on treatment.
- SMS only (Experimental): In addition to standard of care, participants in this arm will receive three SMS reminders. The first SMS will be sent on day one after enrollment into the study. The second SMS will be sent once participant results are ready. If two days after the second SMS the patient has not returned to complete TB diagnosis, a third SMS will be sent. Messages will be automatically sent in either English or Luganda, the commonly spoken local language in the study area. The preferred language of the participant will be determined at enrollment.
  Interventions: Behavioral: SMS
- Phone call only (Experimental): In addition to standard of care, participants in this arm will receive three phone call reminders to complete TB diagnosis. The first phone call will be made on day one after enrollment into the study. The second phone call will be made once participant results are ready. If two days after the second phone call the patient has not returned to complete TB diagnosis, a third phone call will be made. Phone calls will be made in either English or Luganda, the commonly spoken local language in the study area. The preferred language of the participant will be determined at enrollment.
  Interventions: Behavioral: Phone call
- SMS and mobile money incentives (Experimental): In addition to standard of care, participants in this arm will receive three SMS reminders and a transport refund once they complete TB diagnosis. The first SMS will be sent on day one after enrollment into the study. The second SMS will be sent once participant results are ready. If two days after the second SMS the patient has not returned to complete TB diagnosis, a third SMS will be sent. Messages will be automatically sent in either English or Luganda, the commonly spoken local language in the study area. The preferred language of the participant will be determined at enrollment.
  Once participants in this study arm complete TB diagnosis by submitting a sputum sample and collecting back results, a money incentive worth 20,000/= (Twenty thousand shillings only) will be given as a transport refund sent via mobile money.
  Interventions: Behavioral: SMS; Behavioral: Mobile money incentive
- Phone call and mobile money incentives (Experimental): In addition to standard of care, participants in this arm will receive three phone call reminders and a transport refund once they complete TB diagnosis. The first phone call will be made on day one after enrollment into the study. The second phone call will be made once participant results are ready. If two days after the second phone call the patient has not returned to complete TB diagnosis, a third phone call will be made. Phone calls will be made in either English or Luganda, the commonly spoken local language in the study area. The preferred language of the participant will be determined at enrollment.
  Once participants in this study arm complete TB diagnosis by submitting a sputum sample and collecting back results, a money incentive worth 20,000/= (Twenty thousand shillings only) will be given as a transport refund sent via mobile money.
  Interventions: Behavioral: Phone call; Behavioral: Mobile money incentive

INTERVENTIONS:
Behavioral: SMS — Participants in this arm will receive three SMS reminders. The first SMS will be sent on day one after enrollment into the study. The second SMS will be sent once participant results are ready. If two days after the second SMS the patient has not returned to complete TB diagnosis, a third SMS will be sent. Messages will be automatically sent in either English or Luganda, the commonly spoken local language in the study area. The preferred language of the participant will be determined at enrollment.
  Arms: SMS and mobile money incentives; SMS only
Behavioral: Phone call — Participants in this arm will receive three phone call reminders. The first phone call will be made on day one after enrollment into the study. The second phone call will be made once participant results are ready. If two days after the second phone call the patient has not returned to complete TB diagnosis, a third phone call will be made. Phone calls will be made in either English or Luganda, the commonly spoken local language in the study area. The preferred language of the participant will be determined at enrollment.
  Arms: Phone call and mobile money incentives; Phone call only
Behavioral: Mobile money incentive — Once participants in the study arms with mobile money complete TB diagnosis by submitting a sputum sample and collecting back results, a money incentive worth 20,000/= (Twenty thousand shillings only) will be given as a transport refund sent via mobile money.
  Arms: Phone call and mobile money incentives; SMS and mobile money incentives

SUMMARY:
The major challenge in meeting the WHO's End TB Strategy- reducing tuberculosis (TB) deaths by 90% and incidence by 80% is the cascading patient loss-to-follow-up (LTFU) along the continuum of TB care. A systematic review found high levels of pre-treatment LTFU-ranging from 4 to 38%, and was higher in sub-Saharan Africa (18%) compared to Asia (13%). Consequences of pre-diagnosis and pre-treatment LTFU are; untreated TB patients are infectious and can transmit TB to others and not starting TB treatment at all, causes high morbidity and mortality. Therefore, monitoring outcomes of presumptive TB patients is equally important as monitoring treatment outcomes. Short message service (SMS), phone calls and mobile money (MM) incentives have shown promise by improving health outcomes such as uptake of immunization, adherence to TB treatment and antiretroviral therapy (ART). However, there is limited knowledge their effect in increasing linkage to care and treatment for presumptive TB patients in Uganda and sub-Saharan Africa. The aim of this study is therefore to leverage SMS reminders, phone call and MM incentives in improving linkage to care of presumptive TB patients.

This will be a five arm multi-center individual randomized controlled trial implemented in selected high-volume health facilities in Uganda among 1548 presumptive TB patients. The study population will be presumptive TB patients aged 18 years and above identified within the study facilities who do not complete TB diagnosis same day. Completion of TB diagnosis will refer to submitting a sample and obtaining results from the test. Our hypothesis is that using SMS reminders, phone call and Mobile Money incentives will result in increase in the proportion of presumptive TB patients that complete diagnosis and pre-treatment TB cases that initiate treatment.

DETAILED DESCRIPTION:
The major challenge in meeting the WHO's End TB Strategy- reducing TB deaths by 90% and incidence by 80% is the cascading patient loss-to-follow-up (LTFU) along the continuum of TB care. Patients can be lost to follow-up after being identified as presumptive TB cases and never get to test for TB (pre-diagnosis LTFU) or those who test and are confirmed to have TB, can also be lost and never start TB treatment (pre-treatment LTFU). A systematic review found high levels of pre-treatment LTFU-ranging from 4 to 38%, and was higher in sub-Saharan Africa (18%) compared to Asia (13%). Consequences of pre-diagnosis and pre-treatment LTFU are; untreated TB patients are infectious and can transmit TB to others and not starting TB treatment at all, causes high morbidity and mortality. Therefore, monitoring outcomes of presumptive TB patients is equally important as monitoring treatment outcomes. Short message service (SMS), phone calls and mobile money (MM) incentives have shown promise by improving health outcomes such as uptake of immunization, adherence to TB treatment and ART. However, there is limited knowledge their effect in increasing linkage to care and treatment for presumptive TB patients in Uganda and sub-Saharan Africa. The aim of this study is therefore to leverage SMS reminders, phone call and MM incentives in improving linkage to care of presumptive TB patients.

This will be a five arm multi-center individual randomized controlled trial implemented in selected high-volume health facilities in Uganda among 1548 presumptive TB patients. The study population will be presumptive TB patients aged 18 years and above identified within the study facilities who do not complete TB diagnosis same day. Completion of TB diagnosis will refer to submitting a sample and obtaining results from the test.

The study arms will include; i) Standard of care (SOC - control group) ii) SMS only iii) phone call only iv) SMS and MM incentive v) Phone call and MM incentive

Our hypothesis is that using SMS reminders, phone call and Mobile Money incentives will result in increase in the proportion of presumptive TB patients that complete diagnosis and pre-treatment TB cases that initiate treatment.

ELIGIBILITY:
Inclusion Criteria:

* Presumptive TB patient (cough, fever, night sweats, weight loss)
* Requested to have GeneXpert testing
* Aged between 18 and 65 years
* Current resident in the study districts
* Willing to sign informed consent
* Owning a mobile phone
* Able to read

Exclusion Criteria:

* Participant plans to move out of the study area in the next 3 months
* Participation in another related study such as SMS, phone call or mobile money incentive and others

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2355 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Completion of TB diagnosis | 30 days (from being identified as presumptive TB patient)
  This will include completing TB diagnosis using laboratory investigations (GeneXpert) 30 days after being identified as presumptive. This will also include the patient receiving results when ready.
Median time to completing TB diagnosis | Up to 30 days. Determined as Time from when the patient is enrolled on the study to when they complete TB diagnosis
  The time a participant took to complete diagnosis from when they were presumed for TB.

SECONDARY OUTCOMES:
Initiation of TB treatment | 30 days after being confirmed with TB
  This will include initiating treatment within 30 days after being confirmed with TB
Median time to initiating treatment | Up to 30 days. Determined as Time from when the patient is confirmed to have TB to when they initiate TB treatment
  The time a participant took to initiate treatment once confirmed to have TB
Acceptability of the intervention | Through study completion, an average of two months
  This will refer to how acceptable the short message service, phone call and mobile money incentives intervention is in terms of performance, effort, social norms, and facilitating conditions. This will be a post intervention qualitative evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Esther Buregyeya, PhD, Principal Investigator — Makerere University
Locations (5):
- Uganda (5):
  - Luwero General Hospital, Luwero, Kasana
  - Kiruddu National Referral Hospital, Kampala, Makindye
  - Mukono General Hospital, Mukono
  - Entebbe Regional Referral Hospital, Wakiso
  - Wakiso Health Center IV, Wakiso

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be made available to other researchers upon a written request with justification. The study team will review the request and either approve or deny as they deem necessary. Approved requests will only receive patient de-identified data.